CLINICAL TRIAL: NCT01521819
Title: A Pilot, Single-center, Interventional Clinical Trial in Which Subjects With Vascularized Pigment Epithelial Detachment (V-PED) Secondary to AMD With Serous Component Superior to 50% of the Lesion Will Receive Low Voltage Stereotactic Radiotherapy (IRay®) Treatment and Lucentis Treatment as Needed.
Brief Title: Iray for Vascularized Pigment Epithelial Detachment (VPED) Secondary to Age Related Macular Degeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oraya Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLH006
Record Dates: First submitted 2012-01-24; First posted 2012-01-31 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Retinal Pigment Epithelial Detachment With Vascularization; Age Related Macular Degeneration
Keywords: AMD; V-Ped; Vascularized Pigment Epithelial Detachment; Iray; radiation; retina; macula; radiotherapy
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iray plus Lucentis (Experimental): open label arm in which all subjects receive a single 16 gy dose of radiation plus an injection of Lucentis.
  Interventions: Radiation: Iray; Drug: Lucentis

INTERVENTIONS:
Radiation: Iray — The Oraya IRay stereotactic radiotherapy device will be used to deliver a 16 Gy dose of radiation to the macula. The radiotherapy will be delivered in a single session utilizing three sequential beams, each depositing 5.3 Gy at the macula through calculated scleral entry points, crossing the pars plana region of the eye, and overlapping at the same region of the macula.
Drug: Lucentis — Intravitreal injection of Lucentis as needed.

SUMMARY:
This is a pilot, single-center, interventional clinical trial in which subjects will receive 16 Gy of IRay treatment and Lucentis, followed by Lucentis treatment as needed.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of IRay treatment in patients with Vascularized Pigment Epithelial Detachment (V-PED) with serous component superior to 50% of the lesion as determined by decreasing the lesion activity; by decreasing the number of Lucentis injections required during the 12 month study.

ELIGIBILITY:
Inclusion Criteria

* Patients with V-PED with serous component comprising greater than 50% of the lesion area, naïve or previously treated with Lucentis® injections and Photodynamic therapy (PDT) using VisudyneÒ.
* Must have a total lesion size of < 12 disc areas and a lesion with the greatest linear dimension of < 6 mm, but not greater than 3 mm from the center of the fovea to the furthest point on lesion perimeter.
* The distance from the center of the fovea to the nearest edge of the optic disc should be not less than 3 mm. (This distance is confirmed by Oraya software prior to treatment.).
* Must have provided informed consent, documented it in writing, and have been given a copy of the signed informed consent form.
* Must be willing and able to return for scheduled treatment and follow-up examinations for the 1-year duration of the study.
* Must be at least 50 years of age.
* Women must be post-menopausal ≥ 1 year or surgically sterilized, or a pregnancy screen must be performed prior to the study and a reliable form of contraception, approved by the investigator, must be maintained during the study.
* Must have best corrected visual acuity of 75 to 25 letters (inclusive) in the study eye and at least 20 letters in the fellow eye (if both eyes meet all the study criteria, then the eye with the worst vision should be selected as the study eye).

Exclusion Criteria

* CNV due to causes other than AMD, including ocular histoplasmosis syndrome, angioid streaks, multifocal choroiditis, choroidal rupture, or pathologic myopia (spherical equivalent _-8 diopters).
* A globe axial length of < 20 mm or > 26 mm.
* Evidence of diabetes or with retinal findings consistent with diabetic retinopathy or retinopathy for any cause.
* Hypertension that is not controlled with anti-hypertensive medication.
* Prior or concurrent therapies for age related macular degeneration including submacular surgery, subfoveal thermal laser photocoagulation (with or without photographic evidence), or transpupillary thermotherapy (TTT).
* History of radiation to the head in the region of the study eye.
* Previous posterior vitrectomy at any time, YAG capsulotomy or cataract surgery within 3 months, or any other surgery in the study eye within 6 months prior to the screening visit.
* Intravitreal device in the study eye.
* Concomitant disease in the study eye which might interfere with the effect of assessment of the study treatment, including uveitis, acute ocular or periocular infection, retinal vasculopathies (including retinal vein occlusions, etc.) or intraocular pressure > 30 mmHg uncontrollable with medications.
* History of rhegmatogenous retina detachment, optic neuritis or intraocular tumors in the study eye.
* Inadequate pupillary dilation, significant media opacities, or other conditions in the study eye, including cataract, which may interfere with visual acuity or the evaluation of the posterior segment. Subjects likely to need cataract surgery during the 1 year study period should also not be enrolled.
* Known serious allergies to fluorescein dye used in angiography.
* Subjects must not have subretinal hemorrhage or Retinal Pigment Epithelium tear involving the center of the foveal avascular zone.
* Known sensitivity or allergy to Lucentis, or any other drug used in the study, such as topical anesthetic, cycloplegic mydriatics, or lubricating eye gel.
* Contraindication or sensitivity to contact lens application (i.e. corneal dystrophies and recurrent corneal erosions).
* Currently receiving chemotherapy, having completed a course within the 90 days preceding study enrollment, or expecting to begin chemotherapy while participating in the study.
* Current participation in another drug or device clinical trial.
* History of use of drugs with known retinal toxicity, including: chloroquine (Aralen - antimalarial), hydroxychloriquine (Plaquenil - antimalarial), phenothiazines (Thorazine, Stelazine, Mellaril, Prolixin, Trilafon, etc., - tranquilizing antipsychotic medications) and these patients are exhibiting signs of retinal toxicity.
* Concurrent use of systemic anti-VEGF agents.
* Any other condition, which in the judgment of the investigator would prevent the subject from granting consent or completing the study, such as dementia, mental illness (including generalized anxiety disorder, claustrophobia, etc.), or inability to position in the device (due to musculoskeletal problems, etc.).
* History of other significant, uncontrolled disease including cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine or gastrointestinal, metabolic dysfunction, any clinical finding giving reasonable suspicion of a disease or condition that contraindicates the use of intravitreal ranibizumab or that might affect interpretation of the results of the study or render the subject at high risk for treatment complication.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Lesion change as measured with fluorescein angiography. | Baseline and 12 months
  Change in the proportion of the lesion which is active at 12 months.

SECONDARY OUTCOMES:
Number of Lucentis injections | Baseline and 12 months
  Number of Lucentis injections during 12 months
Visual Acuity change | Baseline and 12 months
  Mean change in visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Università Vita-Salute Istituto Scientifico San Raffaele, Milan, Italy